CLINICAL TRIAL: NCT03146819
Title: A Single Time-Point Study to Evaluate the ConforMIS iTotal® (PS) Knee Replacement System Versus Off-the-Shelf Knee Replacement Systems
Brief Title: A Single Time-Point Study to Evaluate the ConforMIS iTotal (PS) Knee Replacement System Versus Off-the-Shelf
Status: Terminated | Type: Observational
Why Stopped: Unable to identify sufficient number of patients to enroll
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: 15-001
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; osteoarthritis knee; total knee replacement; patient specific; total knee arthroplasty; orthopedics
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- iTotal PS KRS: Patients who have had an iTotal (posterior stabilized) knee replacement at least 6 months prior to testing.
  Interventions: Device: iTotal PS Knee Replacement System
- Off-the-Shelf KRS: Patients who have had an off-the-shelf (posterior stabilized) knee replacement at least 6 months prior to testing.
  Interventions: Device: Off-the-Shelf Knee Replacement System

INTERVENTIONS:
Device: iTotal PS Knee Replacement System — Total Knee Replacement systems (Patient Specific)
  Groups: iTotal PS KRS
Device: Off-the-Shelf Knee Replacement System — Total Knee Replacement systems (Off-the-shelf)
  Groups: Off-the-Shelf KRS

SUMMARY:
This study is designed to compare outcome data for patients who have recently undergone surgery with the iTotal® Posterior Stabilizing (PS) Knee Replacement System (hereafter referred to as the "iTotal") versus those who have undergone surgery with Off-the-Shelf (OTS) systems.

DETAILED DESCRIPTION:
This is a prospective, single-time point study that will be conducted in the US.To compare outcomes of these two study groups, this study will include routine office questionnaires such as the Knee Society Score (KSS) and the Knee Injury and Osteoarthritis Outcome Score (KOOS).The functional testing used in this study consists of tests that physical therapists use daily as objective methods to assess patients' functional status. The testing is designed to closely mimic daily activities with which the subjects are familiar.

ELIGIBILITY:
Inclusion Criteria:

* Implant must be a minimum of 6 months post-op and doing well in the opinion of site staff
* Subject has had a knee replacement utilizing a fixed bearing PS (Posterior Stabilized) implant design
* > 18 years of age
* Willingness to participate in the clinical study, to give informed consent, and to perform all evaluations

Exclusion Criteria:

* Simultaneous or staged bilateral procedure
* BMI > 40
* Other physical disability that requires an aid for walking or disability affecting the hips, spine, contralateral knee or other joint that limits function
* Participation in another clinical study which would confound results
* Inability to complete the protocol in the opinion of the clinical staff due to safety or other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include a 1:1 ratio of patients enrolled into both the iTotal arm and the off-the-shelf total knee arm.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Functional testing differences | At least 6 months post-surgery
  Physical therapy functional testing between the iTotal PS and off-the-shelf PS implants

SECONDARY OUTCOMES:
Knee Society Clinical Rating Score | At least 6 months post-surgery
  Comparison of scores and sub-scores from the following questionnaires between the study arms
The Knee Injury and Osteoarthritis Outcome Score (KOOS) | At least 6 months post-surgery
  Comparison of scores and sub-scores from the following questionnaires between the study arms

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cannova, MD, Principal Investigator — Bethesda Orthopedic
Locations (1):
- Bethesda Orthopedic, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bourne RB, Chesworth BM, Davis AM, Mahomed NN, Charron KD. Patient satisfaction after total knee arthroplasty: who is satisfied and who is not? Clin Orthop Relat Res. 2010 Jan;468(1):57-63. doi: 10.1007/s11999-009-1119-9. PMID 19844772
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Lepage C, Noreau L, Bernard PM. Association between characteristics of locomotion and accomplishment of life habits in children with cerebral palsy. Phys Ther. 1998 May;78(5):458-69. doi: 10.1093/ptj/78.5.458. PMID 9597060
- [Background] McCarthy CJ, Oldham JA. The reliability, validity and responsiveness of an aggregated locomotor function (ALF) score in patients with osteoarthritis of the knee. Rheumatology (Oxford). 2004 Apr;43(4):514-7. doi: 10.1093/rheumatology/keh081. Epub 2004 Jan 13. PMID 14722348
- [Background] Mizner RL, Petterson SC, Clements KE, Zeni JA Jr, Irrgang JJ, Snyder-Mackler L. Measuring functional improvement after total knee arthroplasty requires both performance-based and patient-report assessments: a longitudinal analysis of outcomes. J Arthroplasty. 2011 Aug;26(5):728-37. doi: 10.1016/j.arth.2010.06.004. Epub 2010 Sep 20. PMID 20851566
- [Background] Noble PC, Conditt MA, Cook KF, Mathis KB. The John Insall Award: Patient expectations affect satisfaction with total knee arthroplasty. Clin Orthop Relat Res. 2006 Nov;452:35-43. doi: 10.1097/01.blo.0000238825.63648.1e. PMID 16967035
- [Background] Nordin E, Rosendahl E, Lundin-Olsson L. Timed "Up & Go" test: reliability in older people dependent in activities of daily living--focus on cognitive state. Phys Ther. 2006 May;86(5):646-55. PMID 16649889
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Suda AJ, Seeger JB, Bitsch RG, Krueger M, Clarius M. Are patients' expectations of hip and knee arthroplasty fulfilled? A prospective study of 130 patients. Orthopedics. 2010 Feb;33(2):76-80. doi: 10.3928/01477447-20100104-07. PMID 20192137
- [Background] Wall JC, Bell C, Campbell S, Davis J. The Timed Get-up-and-Go test revisited: measurement of the component tasks. J Rehabil Res Dev. 2000 Jan-Feb;37(1):109-13. PMID 10847578
- [Background] Zaino CA, Marchese VG, Westcott SL. Timed up and down stairs test: preliminary reliability and validity of a new measure of functional mobility. Pediatr Phys Ther. 2004 Summer;16(2):90-8. doi: 10.1097/01.PEP.0000127564.08922.6A. PMID 17057533